CLINICAL TRIAL: NCT01769482
Title: Understanding of Chest Pain in Microvascular Disease Proved by Cardiac Magnetic Resonance Image
Acronym: UMPIRE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-07-048
Record Dates: First submitted 2012-11-20; First posted 2013-01-16 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2012-11

CONDITIONS: Microvascular Angina
Keywords: microvascular angina; PDE-5 inhibitors; Heart disease; Ischemia; Cardiac MRI
MeSH Terms: conditions — Microvascular Angina; Heart Diseases; Ischemia | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Udenafil (Experimental): 70 subjects will undergo baseline testing and then be randomized into a clinical parallel trial of udenafil 100mg or placebo po q d for 3 months.
  Interventions: Drug: Udenafil
- Placebo (Placebo Comparator): 70 subjects will undergo baseline testing and then be randomized into a clinical parallel trial of udenafil 100mg or placebo po q d for 3 months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Udenafil — 70 subjects will undergo baseline testing and then be randomized into a clinical parallel trial of udenafil 100mg po q d for 3 months.
  Other Names: Zydena
  Arms: Udenafil
Drug: placebo
  Arms: Placebo

SUMMARY:
Current therapeutic options for a well-recognized group of patients with anginal symptoms-a positive exercise tolerance testing, SPECT or perfusion defect in MRI but angiographically normal coronary arteries-are limited. The condition, referred to as microvascular angina (MVA) or cardiac syndrome X, is not as benign as originally reported-patients presenting with unstable angina and nonobstructive atherosclerotic coronary artery disease have a 2% risk of death or myocardial infarction at 30 days of follow-up. It is more common in women in whom the first presentation of angina occurs either perimenopausally or postmenopausally. Aberrant flow-mediated coronary vasomotion is pivotal in the pathogenesis (systemic) impairment in endothelial function. Indeed, some centers use systemic assessments of vascular function in their diagnostic pathways for this group of women. It was recently suggested that endothelial dysfunction may lead to myocardial ischemia.

In the present study, the investigators tested the hypothesis that udenafil offers dual benefits of improving vascular function and lessening ischemia in women with angina, perfusion defect in cardiac MRI, and normal coronary arteries.

DETAILED DESCRIPTION:
The aim of this study is that udenafil offers dual benefits of improving vascular function and lessening ischemia in women with microvascular angina, perfusion defect in cardiac MRI, and normal coronary arteries.

The UMPIRE trial is a multi-center, prospective, randomized, placebo controlled trial, designed to evaluate the effect of udenafil in improvement of myocardial stress perfusion defect in cardiac MRI, in women patients with microvascular angina. A total of 70 patients will be randomized to udenafil(100 mg q d) or placebo treatment. The primary end point of the study is Change of perfusion defect over 25% of baseline defect in adenosine-stress cardiac MRI after 3-month treatment. The secondary endpoints of this study are change of perfusion defect less than 25% of baseline defect in adenosine-stress cardiac MRI after 3-month treatment, decrement of frequency of chest pain, improvement of ST-depression in stress test, improvement of duke score in stress test, improvement of QoL assessment by SF-36 questionnaire, improvement of sexual dysfunction assessment by BISF-W self-questionnaire and improvement of biomarkers foe endothelial function.

ELIGIBILITY:
Inclusion Criteria:

1. MVA patients with typical symptom and positive adenosine-stress cardiac MRI and with normal coronary artery in coronary angiogram or coronary artery CT angiography.
2. Definition of positive adenosine-stress MRI: perfusion defect > 25% of transmurality ( by 2 radiologist based on visual assessment and qualitative assessment in core-lab)
3. Gender: female
4. Age: 18-80

Exclusion Criteria:

1. The patient with contraindication to MR contrast media or MR Imaging
2. LVEF < 50%
3. Any heart rhythm abnormality other than sinus rhythm
4. Valvular heart disease with more than moderate degree
5. Renal failure
6. Congestive Heart Failure
7. Myocardial infraction
8. Myocarditis
9. Congenital heart disease
10. Pericarditis
11. Variant angina (positive provocation test with Ergonovine or acetylcholine)
12. GERD (conformed by esophagogastroduodenoscopy)
13. Pregnant women with suspected, pregnant women or women with lactation
14. QT prolongation syndrome or take drugs that prolong the QT interval - Antiarrhythmics class IA; quinidine, procainamide - Antiarrhythmics class III; amiodarone, sotalol
15. Preanalytical within 30 days of screening in a clinical trial that may affect the influence of udenafil

    - Other PDE5 inhibitors (ex. Sildenafil, tadalafil)

    - Nitrates/ NO donor (ex. Nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, amyl nitrate/nitrite, sodium nitroprusside, nicorandil)
16. Preanalytical within 7 days of screening in a clinical trial that may affect the metabolism of udenafil

    * Antibacterials (ex. Erythromycin)
    * Antifungals (ex. Itraconazole, ketoconazole)
    * Antivirals (ex. Ritonavir, saquinavir, amprenavir, indinavir, nelfinavir)
    * Cimetidine
    * Grapefruit juice
17. Allergy or sensitivity with PDE 5 inhibitors

    -

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
to change of perfusion defect over 25% of baseline defect in adenosine-stress cardiac MRI after 3-month treatment. | baseline, 3 months after treatment

SECONDARY OUTCOMES:
to change of perfusion defect less than 25% of baseline defect in adenosine-stress cardiac MRI after 3-month treatment | baseline, 3 months after treatment

OTHER OUTCOMES:
to change of frequency of chest pain | baseline, 3 months after treatment
to change of improvement of ST-depression in ECG | baseline, 3 months after treatment
to change of QoL(Quality of Life) | baseline, 3 months after treatment
to change of sexual dysfunction | baseline, 3 months after treatment
to change of improvement of biomarkers for endothelial function | baseline and 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Ji Park, M.D.,Ph.D., Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Guro Hospital, Seoul

REFERENCES:
- [Derived] Park SJ, Park JJ, Choi DJ, Chun EJ, Choi SI, Kim SM, Jang SY, Ahn S, Choe YH. Understanding of chest pain in microvascular disease proved by cardiac magnetic resonance image (UMPIRE): study protocol for a randomized controlled trial. Trials. 2014 Aug 26;15:333. doi: 10.1186/1745-6215-15-333. PMID 25154607